CLINICAL TRIAL: NCT06465966
Title: UFPTI 2403-PR12: Real-Time Volumetric Ionizing Radiation Acoustic Imaging for In-vivo Proton Treatment Monitoring in Pencil-Beam Scanning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202400573
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iRAI data collection (Experimental): Radiation therapists will position the participant on the treatment table. After the participant is setup, a water bag will be placed on his abdomen and a 2D transducer is placed on top of the water bag. The 2D transducer is held in place by an articulated arm attached to the treatment table. The water bag serves as a path for the photo acoustic waves created during treatment to be detected by the 2D transducer and captured for data collection.
  Interventions: Device: iRAI

INTERVENTIONS:
Device: iRAI — Ionizing-radiation photo acoustic imaging (iRAI) is a method of collecting images from inside the body using acoustic (sound) waves. Researchers will collect iRAI during a participant's radiation treatments. Researchers will use this imaging to examine the delivery and dose of the radiation to the participant's prostate. Researchers will also compare the delivery and dose calculated from iRAI to the expected doses that were calculated from CT images which are done as standard of care.

SUMMARY:
The purpose of this study is to evaluate the use of ionizing-radiation photo acoustic imaging (iRAI) for proton radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Disease: Prostate cancer
* Treatment site:
* Prostate or prostate and seminal vesicle
* No regional lymph node is involved
* Patient's body weight: Patient's body weight is less than 350 lbs to consider the total weight limit that the ProteusONE treatment table and the robotic arm can operate
* Treatment volume size: maximum size less than 15 x 15 cm in a cross-section and a thickness less than 20 cm to consider 2D transducer matrix size
* Provision to sign the consent form and understand the non-invasiveness of iRAI
* Patient agreement on tolerance on placing a water bag to acquire iRAI during treatment
* Treatment modality: Proton radiation therapy with UFHPTI's ProteusONE gantry using PBS

Exclusion Criteria:

* A patient who would not be tolerable or will feel nervous about being touched on the skin with a water bag
* A patient with a significant medical implant or hardware in the treatment area

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Proton treatment dose overlay between predicted values and iRAI in CT images at the center plane of a tumor to achieve | Approximately 36 months for trial accrual
  95% confidence interval in the gamma passing rate higher than 90% using 5%/5 mm criteria

SECONDARY OUTCOMES:
Reliability of range discrepancies between predicted values and iRAI during 3-day treatments at the proximal, center, and distal plane of a tumor to achieve | Approximately 36 months for trial accrual
  Standard error of less than 5% between the passing rates when using a 5 mm distance-to-agreement

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Florida Health Proton Therapy Institute, Jacksonville, Florida, United States